CLINICAL TRIAL: NCT06992427
Title: High-Dose Prophylactic Gabapentin (HOPE) to Prevent Opioid Use for Oral Mucositis Pain During Head and Neck Chemoradiotherapy: A Phase III Clinical Trial
Brief Title: High-dose Prophylactic Gabapentin (HOPE) vs. Placebo to Prevent Opioid Use for Oral Mucositis Pain During Concurrent Chemoradiation for Head and Neck Cancer
Acronym: HOPE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: A222301; NCI-2025-00501 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2025-04-28; First posted 2025-05-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Stage I Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage II Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage III Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage IV Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Gabapentin; Radiotherapy; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Placebo) (Placebo Comparator): Starting by radiation treatment 8, patients receive placebo PO QD on day 1, BID on day 2, then TID starting day 3 onward. Patients also receive standard of care radiation, chemotherapy and pain medications. Treatment with placebo continues in the absence of disease progression or unacceptable toxicity, until the symptoms of oral mucositis and other treatment effects begin to resolve and other pain medications has been stopped. Patients then continue to receive placebo TID for 9 additional days, at sequentially smaller doses, then BID for 1 day and QD for one day before stopping. Patients undergo blood sample collection throughout the study.
  Interventions: Drug: Placebo; Drug: Chemotheraphy; Radiation: Radiation Therapy; Drug: Analgesic Agent; Procedure: Biospecimen Collection; Other: Survey Administration
- Arm II (Gabapentin) (Experimental): Starting by radiation treatment 8, patients receive gabapentin PO QD on day 1, BID on day 2, then TID starting day 3 onward. Patients also receive standard of care radiation, chemotherapy and pain medications. Treatment with gabapentin continues in the absence of disease progression or unacceptable toxicity, until the symptoms of oral mucositis and other treatment effects begin to resolve and other pain medications has been stopped. Patients then continue to receive gabapentin TID for 9 additional days, at sequentially smaller doses, then BID for 1 day and QD for one day before stopping. Patients undergo blood sample collection throughout the study.
  Interventions: Drug: Gabapentin; Drug: Chemotheraphy; Radiation: Radiation Therapy; Drug: Analgesic Agent; Procedure: Biospecimen Collection; Other: Survey Administration

INTERVENTIONS:
Drug: Gabapentin — Given PO
  Other Names: Gralise; Neurontin
  Arms: Arm II (Gabapentin)
Drug: Placebo — Given PO
  Arms: Arm I (Placebo)
Drug: Chemotheraphy — Receive standard of care chemotherapy
Radiation: Radiation Therapy — Undergo standard of care radiation
Drug: Analgesic Agent — Receive standard of care pain medication
Procedure: Biospecimen Collection — Undergo blood sample collection
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase III trial tests if gabapentin can prevent the need for opiate pain medication for mouth sores (oral mucositis) in patients undergoing treatment with chemotherapy and radiation for squamous cell carcinoma of the head and neck region. Oral mucositis is a common side effect of radiation treatment and can cause severe pain, dysphagia, and weight loss resulting in feeding tube placement, worse health-related quality of life, treatment interruptions, unplanned hospitalizations, and significant financial burden. Mucositis pain is often treated with opioid pain medications which do provide pain relief but have many known side effects not limited to mental clouding, constipation, fatigue, endocrinopathy, neurotoxicity, sleep-disordered breathing, and most distressingly persistent opioid use. Gabapentin may help relieve pain from oral mucositis caused by radiation while also reducing the need for opiate pain medications for patients receiving chemotherapy and radiation for squamous cell carcinoma of the head and neck region

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether prophylactic high dose gabapentin, titrated to a dose of 3600 mg (1200 mg three times per day [TID]), is superior to placebo in increasing the proportion of patients not needing opiates while undergoing chemoradiation therapy.

SECONDARY OBJECTIVES:

I. To determine whether prophylactic high dose gabapentin is superior to placebo in prolonging the time to first opioid use while undergoing chemoradiation therapy.

II. To determine whether prophylactic high dose gabapentin is superior to placebo in improving patient reported pain scores using the 0-10 numerical rating scale (NRS) from baseline to 4 weeks after the end of chemoradiation therapy.

EXPLORATORY OBJECTIVES:

I. To explore the duration of opioid use from the time of initiation to cessation by arm as well as describe the proportion of patients remaining on opioids at 3 months, 6 months, and 1 year by arm.

II. To explore the trajectory of patient reported symptom and quality of life outcomes using the Oral Mucositis Weekly Questionnaire (OMWQ) by arm.

III. To explore the trajectory of patient reported symptom and quality of life outcomes using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-30 (EORTC QLQ-30) by arm.

IV. To explore the trajectory of patient reported symptom and quality of life outcomes using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck-43 (EORTC QLQ-H&N43) by arm.

V. To evaluate the adverse event profiles of prophylactic high dose gabapentin versus placebo.

VI. To assess the tolerance of high dose gabapentin. VII. To explore the trajectory of patient health using patient body mass index (BMI) and creatinine, absolute neutrophil count (ANC) as routinely obtained by arm.

VIII. To describe the incidence of feeding tube requirement during and after chemoradiation therapy by arm.

IX. To describe the dose of prescribed opioids standardized using the Morphine Milligram Equivalent calculator by arm.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Starting by radiation treatment 8, patients receive placebo orally (PO) once daily (QD) on day 1, twice daily (BID) on day 2, then three times daily (TID) starting day 3 onward. Patients also receive standard of care radiation, chemotherapy and pain medications. Treatment with placebo continues in the absence of disease progression or unacceptable toxicity, until the symptoms of oral mucositis and other treatment effects begin to resolve and other pain medications has been stopped. Patients then continue to receive placebo TID for 9 additional days, at sequentially smaller doses, then BID for 1 day and QD for one day before stopping. Patients undergo blood sample collection throughout the study.

ARM II: Starting by radiation treatment 8, patients receive gabapentin PO QD on day 1, BID on day 2, then TID starting day 3 onward. Patients also receive standard of care radiation, chemotherapy and pain medications. Treatment with gabapentin continues in the absence of disease progression or unacceptable toxicity, until the symptoms of oral mucositis and other treatment effects begin to resolve and other pain medications has been stopped. Patients then continue to receive gabapentin TID for 9 additional days, at sequentially smaller doses, then BID for 1 day and QD for one day before stopping. Patients undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 4 weeks, 3 months and 6 months after the last dose of chemoradiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of disease: Squamous cell carcinoma of the head and neck region.

  * Stage: I-IV
* No prior treatment for head and neck cancer
* Planned treatment with cisplatin-based chemoradiation therapy (weekly or once every 3 weeks [q 3 week])
* Able to swallow capsules whole
* No known hypersensitivity to gabapentin or its ingredients
* No patients on dialysis or with transplanted organs
* No prior surgery or radiation for head and neck cancer and/or are being treated for recurrent head and neck cancer. Patients with a history of surgery and radioactive iodine for the treatment of thyroid cancer are eligible. Concurrent cancer therapy for other cancers is not allowed
* No planned surgery or chemotherapy or immunotherapy following 7 weeks of standard chemoradiation treatment
* No known brain metastases
* No nonprescribed use of any opioids (including heroin) within 6 months prior to registration
* No prescribed medications for chronic and/or long-term pain and/or neuropathy, including patients under treatment of a pain specialist or substance abuse programs. Acute post-biopsy medications are allowed if the patient has discontinued them 3 days prior to study registration
* No current treatment with mefloquine
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Creatinine ≤ 1.5 x upper limit of normal (ULN)
* Not pregnant and not nursing, because this study involves both radiation and chemotherapy. In addition, the genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown. Therefore, for women of childbearing potential, a negative pregnancy test done < 7 days prior to registration is required. Women must agree to using contraception for the duration of receiving study drugs and for 6 months after completing chemoradiation
* Not taking medications for a psychotic psychiatric illness
* No existing diagnosis of sleep apnea
* No acute narrow-angle glaucoma
* No uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No investigational agent within 30 days prior to registration
* No enrollment on other studies of systemic pain control agents
* Language: In order to complete the mandatory patient-completed measures, participants must be able to speak and read English or Spanish
* Patients with impaired decision making are not eligible for study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2029-08-15 (Estimated); Study Completion 2031-04-15 (Estimated)

PRIMARY OUTCOMES:
Need to use opioids during chemoradiation therapy (CRT) | Up to 7 weeks
  Will be tested using a two-sample test of proportions. Will report the proportion of patients not using opioids within the 7 weeks of CRT in the two arms and the 95% confidence interval (CI) of the difference in the proportions.

SECONDARY OUTCOMES:
Time to first opioid use | Up to 9 weeks
  Time to first opioid use, defined as the time from randomization to the first occurrence of opioid use during CRT, censoring patients alive and opioid free at CRT completion. Death or disease progression before first opioid use during CRT will be treated as competing events. Cumulative incidence functions will be used to estimate the percentage of patients who experience the competing events within the arms. Differences between the cumulative incidence functions between the arms will be tested for statistical significance using the procedure of Gray. The cumulative incidence percentage at the end of CRT by arm will be reported.
Patient-reported pain scores | Through 4 weeks post CRT (up to 14 weeks)
  Pain score responses of question #5 on the Oral Mucositis Weekly Questionnaire-Head and Neck Cancer (OMWQ-HN) survey at each collected timepoint for each arm. This NRS item asks a respondent to rate their overall mouth and throat soreness during the past week from 0 (no soreness) to 10 (worst possible soreness). Will apply longitudinal modeling of the patient-reported pain scores through four weeks post CRT treatment. Will report each time-specific comparison between arms with a 95% CI.

OTHER OUTCOMES:
Need to use opioids during CRT by sex | Up to 7 weeks
  Will be assessed between arms and the corresponding 95% CIs will be provided by sex (male; female).
Need to use opioids during CRT by race | Up to 7 weeks
  Will be assessed between arms and the corresponding 95% CIs will be provided by race (white; other).
Need to use opioids during CRT by ethnicity | Up to 7 weeks
  Will be assessed between arms and the corresponding 95% CIs will be provided by ethnicity (Not Hispanic or Latino; Hispanic or Latino).
Duration of opioid use | Though 4 weeks post CRT (up to 14 weeks)
  Will report the number of patients and descriptively summarize the duration of opioid use from the time of initiation to cessation, or 4 weeks post-CRT (acute opioid use), whichever comes first. Descriptive statistics will include the mean, standard deviation, median, interquartile range, minimum, and maximum.
Global health | Through 4 weeks post CRT (up to 14 weeks)
  Measured via OMWQ-HN. The first two items of the OMWQ-HN assess global health and quality of life and are rated on a seven-point scale, with one indicating very poor and seven indicating excellent. The focus will be on the interaction effect, which concerns comparisons of the patterns of changes in the mean patient-reported pain scores. In addition to plotting the model-based mean response profiles by arm, will report each time specific comparison between arms with a 95% CI.
Patient reported oral mucositis symptoms. | Through 4 weeks post CRT (up to 14 weeks)
  Measured via OMWQ-HN. The third item of the OMWQ-HN assesses mouth and throat soreness and is rated on a five-point scale, with zero indicating no soreness and four indicating extreme soreness. The focus will be on the interaction effect, which concerns comparisons of the patterns of changes in the mean patient-reported pain scores. In addition to plotting the model-based mean response profiles by arm, will report each time specific comparison between arms with a 95% CI.
Mouth and throat soreness | Through 4 weeks post CRT (up to 14 weeks)
  Measured via OMWQ-HN. The last three items of the OMWQ-HN assess the degree of mouth and throat pain and soreness using an 11-point scale, with zero indicating no pain or soreness and 10 indicating the worst pain or soreness imaginable or possible. The focus will be on the interaction effect, which concerns comparisons of the patterns of changes in the mean patient-reported pain scores. In addition to plotting the model-based mean response profiles by arm, will report each time specific comparison between arms with a 95% CI.
Impact of mouth and throat soreness on patient function | Through 4 weeks post CRT (up to 14 weeks)
  Measured via OMWQ-HN. The fourth item of the OMWQ-HN, which is made up six different activities each rated on a five-point scale (0 = not limited and 4 = unable to do), assesses the impact of mouth and throat soreness on patient function; responses to the six different activities are summed (range: 0 to 24), with lower scores being better. The focus will be on the interaction effect, which concerns comparisons of the patterns of changes in the mean patient-reported pain scores. In addition to plotting the model-based mean response profiles by arm, will report each time specific comparison between arms with a 95% CI.
Incidence of symptoms or problems | Through 4 weeks post CRT (up to 14 weeks)
  Measured on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck-43. The scales and singles arms range from 0-100, with higher scores indicating fewer symptoms or problems; a change of 10 units on the 0-100 response scale is regarded as considered clinically important. The focus will be on the interaction effect, which concerns comparisons of the patterns of changes in the mean patient-reported pain scores. In addition to plotting the model-based mean response profiles by arm, will report each time specific comparison between arms with a 95% CI.
Incidence of adverse events (AE) | Up to approximately 2 years
  As scored using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v 5.0). Will be summarized within arms by reporting the number and percentages of patients. Specifically, to evaluate the AE profiles within each arm, the maximum grade for each type of AE will be recorded for each patient and frequency tables will be reviewed to determine overall patterns; additionally, the proportion of somnolence, confusion, and gait disturbance using NCI CTCAE v 5.0 will be estimated within arms with the exact 90% CI.
Tolerance of gabapentin | Up to the 9 weeks
  Defined as ≥ 80% adherence (yes; no) to gabapentin during CRT. The proportion of patients that complete CRT and tolerate gabapentin during CRT will be reported.
Body mass index | Up to the 9 weeks
  Descriptive statistics will include the mean, standard deviation, median, interquartile range, minimum, and maximum.
Creatinine | Up to the 9 weeks
  Descriptive statistics will include the mean, standard deviation, median, interquartile range, minimum, and maximum.
Absolute neutrophil count | From baseline to the completion of CRT
  Descriptive statistics will include the mean, standard deviation, median, interquartile range, minimum, and maximum.
Dose of prescribed opioids | Up to 7 weeks.
  The patient average dose of prescribed opioids will be standardized using the Morphine Milligram Equivalent calculator. Will summarize the within patient average dose of prescribed opioids according to arm using the mean, standard deviation, median, interquartile range, minimum, and maximum values.
Incidence of Feeding Tube | Through 4 weeks post CRT (up to 14 weeks)
  Will report the frequency and percentage of patients within each arm who require a feeding tube during CRT.

CONTACTS AND LOCATIONS:
Locations (150):
- United States (150):
  - Arizona Center for Cancer Care - Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Arizona Center for Cancer Care - Biltmore, Phoenix, Arizona
  - Arizona Center for Cancer Care - Phoenix, Phoenix, Arizona
  - Arizona Center for Cancer Care - Osborn, Scottsdale, Arizona
  - Arizona Center for Cancer Care - Scottsdale, Scottsdale, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - Arizona Center for Cancer Care, Tempe, Arizona
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health Physicians Partners Radiation Medicine at Queens, Forest Hills, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Queens Cancer Center, Rego Park, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Aultman Health Foundation, Canton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided